CLINICAL TRIAL: NCT01938586
Title: Comparison of Traditional Superficial Cutaneous Sutures Versus Steri-Strip Coaptive Film in Layered Dermatologic Closures on the Back - a Prospective, Randomized, Split-scar Study
Brief Title: Comparison of Traditional Superficial Cutaneous Sutures Versus Steri-Strip Coaptive Film in Layered Dermatologic Closures
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Director of Cosmetic Dermatology, Vice-Chair of Operations, Henry Ford Health System
Other Study IDs: SYDO-2013
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2013-09

CONDITIONS: Wound Cosmesis
Keywords: Scar; Appearance
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Surgical excision
  Interventions: Other: Steri-Strip; Other: Superficial sutures

INTERVENTIONS:
Other: Steri-Strip
Other: Superficial sutures

SUMMARY:
The purpose of this study is to compare the cosmetic outcome between buried intradermal and superficial cutaneous suture closures versus buried intradermal sutureand superficial Steri-Strip closures in the bilayered repair of dermatologic wounds on the back following elliptical excision of benign or malignant lesions

ELIGIBILITY:
Inclusion Criteria:

* 18 years or greater in age
* Simple excision of benign or malignant lesion on the back
* Final scar length of at least 3cm

Exclusion Criteria:

* Known history of keloid formation or hypertrophic scars
* Known adhesive allergy
* Pregnancy or active breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient dermatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Overall scar appearance as evaluated by the Patient and Observer Scar Assessment Scale | 6 months

SECONDARY OUTCOMES:
Rates of postoperative complications | 6 months
  Assessment of scar erythema, swelling, infection, drainage, dehiscence
Time for closure of each split half portion of wound | 1 hour (intraoperative)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Dermatology Clinic, Detroit, Michigan, United States